CLINICAL TRIAL: NCT06640725
Title: A Phase II Study of TPEx (Taxotere-platinum-cetuximab) Followed by a Maintenance With Avelumab and Cetuximab in First Line Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (TATIANA)
Brief Title: Study of TPEx Followed by a Maintenance With Avelumab and Cetuximab in First Line Recurrent or Metastatic Squamous Cell Carcinoma of the H&N
Acronym: TATIANA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2024-01; 2023-510559-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Recurrence | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPEx-Avelumab-Cetuximab (Experimental): Induction (TPEx regimen: up to 4 cycles Q3W) Cisplatin 75 mg/m² or Carboplatin AUC 5 every 3 weeks (±2 days). Docetaxel 75 mg/m² every 3 weeks (±2 days). Cetuximab with a loading dose of 400mg/m² at C1D1 and after 250mg/m² every week (±2 days).
  Cetuximab 500 mg/m² every 2 weeks (±3 days) (according to current recommendations [35]) Avelumab 10 mg/kg every 2 weeks (±3 days)
  Interventions: Drug: Avelumab administration at 10mg/kg; Drug: Cetuximab (Erbitux)

INTERVENTIONS:
Drug: Avelumab administration at 10mg/kg — Maintenance (until progression, unacceptable toxicity or if CR > 1 year, as per investigator choice)
  Avelumab 10 mg/kg every 2 weeks (±3 days)
Drug: Cetuximab (Erbitux) — Maintenance (until progression, unacceptable toxicity or if CR > 1 year, as per investigator choice)
  Cetuximab 500 mg/m² every 2 weeks (±3 days) (according to current recommendations [35])

SUMMARY:
The main objective of this research is to increase the life expectancy of patients with advanced mouth and throat cancer, by adding avelumab to the standard TPEx treatment.

All participants in this research will receive the same treatment which will take place in two phases:

* 1st phase chemotherapy + immunotherapy: standard reference treatment (Docetaxel + cisplatin or carboplatin + cetuximab)
* 2nd phase immunotherapy: cetuximab combined with avelumab which is the treatment under study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women ≥ 18 years and < 75 years.
2. Histologically confirmed recurrent and/or metastatic SCCHN (oral cavity, pharynx, larynx), not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy); squamous cell carcinoma of unknown primary if HPV positive.
3. Detection of PD-L1 protein expression in formalin-fixed, paraffin-embedded (FFPE) SCCHN tissue samples determined by Combined Positive Score (CPS) ≥1 using local IHC assay.
4. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
5. Patients without contra indication to TPEx (either with cisplatin or carboplatin), to docetaxel, cetuximab and to immunotherapy (avelumab).Investigators must refer to the last updated version of Summary of product Characteristics (SPC) of the products.
6. Documentation of p16 status as surrogate of human papillomavirus (HPV) status of tumor for SCC of the oropharynx.
7. Measurable disease by CT or MRI per RECIST 1.1 criteria.
8. In case of radiotherapy given without systemic treatment, prior curative radiation therapy must have been completed at least 4 weeks before TPEx administration and/or prior palliative radiotherapy must have been completed at least 2 weeks before TPEx administration.
9. Screening laboratory values must meet the following criteria (using NCI-CTCAE v5) and should be obtained within 14 days prior to eligibility check:

   1. WBC > 2000/μL
   2. Polynuclear neutrophils >1.5 x 109/L
   3. Platelets > 100 x 109/L
   4. Hemoglobin > 9.0 g/mL
   5. ALAT/ASAT< 3.0 x ULN in the absence of liver metastases or < 5x ULN in the presence of liver metastases
   6. Bilirubin < 1.5 x ULN (except Gilbert Syndrome: < 3.0 mg/dL)
   7. Creatinine clearance > 60 mL/min (measured or calculated by preferably Cockcroft and Gault formula) for cisplatin administration and creatinine clearance between ≥ 40 mL/min and ≤ 60 mL/min (measured or calculated by preferably Cockcroft and Gault formula) for carboplatin administration.
10. Calcium levels must be normalized and maintained within normal limits for study entry. Medical management of calcium levels is permitted. Note: Normal calcium levels may be based on ionized calcium or adjusted for albumin.
11. Recovery to baseline or ≤ Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5 from AE(s) related to any prior treatments unless AE(s) are deemed clinically non-significant by the Investigator and/or stable on supportive therapy.
12. Women of childbearing potential must have a negative serum or urine pregnancy test at the eligibility check. The pregnancy test must be done within 72 hours before eligibility check.
13. Both men and women (of childbearing potential) who are sexually active must agree to use highly effective contraceptive method(s) from ICF signature to at least 7 months post-treatment for women and 4 months post-treatment for men.

Exclusion Criteria:

* 1.Prior systemic chemotherapy for the head and neck carcinoma, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to study entry.

  2.Histologically confirmed recurrent or metastatic carcinomas of the nasopharynx, squamous cell carcinoma of unknown HPV negative primary, or salivary gland or non-squamous histologies (e.g., mucosal melanoma) are not allowed.

  3.Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.

  4.Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

  5.Subjects with active, known or suspected autoimmune disease. Subjects with stabilized type I diabetes mellitus under treatment, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

  6.Subjects with a condition requiring systemic chronic administration of corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of eligibility check. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

  7.Patients having received prior therapy with anti-PD1, anti-PD-L1(or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).

  8.Prior anti-EGFR treatment received less than 6 months before eligibility check.

  9.Patients with known positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

  10.Patients with known positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.

  11.Use of non-oncology vaccines containing live virus or bacteria for prevention of infectious diseases within 4 weeks prior to eligibility check. The use of the inactivated seasonal influenza vaccine is allowed.

  12.History of severe hypersensitivity reaction to any human monoclonal antibody.

  13.Severe concurrent psychiatric conditions that would limit compliance with study requirements.

  14.Serious systemic infection requiring hospital treatment with intravenous antibiotics within 14 days prior eligibility check.

  15.History of organ transplant. 16.Patients presenting hemorrhagic tumor, only if carboplatin is administrated. 17.Concomitant phenytoin and fosphenytoin medication during the study treatment period.

  18.History of allergy to red meat or tick bites or positive results of tests for IgE antibodies against cetuximab (α-1-3-galactose).

  19.Interstitial lung disease. 20. History of uncontrolled or symptomatic cardiac disease. 21. Individual deprived of liberty by judicial or administrative decision, or under any kind of guardianship.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-10-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1, 2and 3 years
  Overall survival (OS) defined as the time from the inclusion in the study to death due to any cause or the last follow-up contact for patients who are alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No
IPD contains personal data